CLINICAL TRIAL: NCT07000435
Title: Assessing Thickness Changes Following the Use of 3D-Printed Vs. Custom-Made Mouth Guards to Prevent Traumatic Dental Injuries in Children Practicing Contact Sports: A Randomized Clinical Trial.
Brief Title: Comparative Assessment of Thickness Changes in 3D-Printed vs. Custom-Made Mouth Guards for Children in Contact Sports
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Tawfik Mohamed, Master's Candidate, Department of Pediatric Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Thickness of Mouthguards
Record Dates: First submitted 2025-05-24; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Mouthguard Use Orofacial Injuries Prevention 3D Printed Mouthguard Traditional Custom-made Mouthguard Occlusal Thickness Changes
Keywords: 3D printed mouthguard traditional custom-made mouthguard occlusal thickness CAD/CAM 3D printer Children Pediatric Dentistry Contact sports thickness changes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two groups: one group will receive traditional custom-made mouthguards, and the other will receive 3D-printed custom-made mouthguards. Each participant will remain in their assigned group throughout the study period, and outcomes will be assessed independently for each group.
Who Masked: Participant, Investigator
Masking Description: Blinding will be applied at multiple levels to minimize bias in this study. Since both the traditional custom-made and 3D-printed mouthguards have a similar appearance, this study will be double-blinded to both the principal investigator and the patients in each study group, thereby reducing expectation bias. A coach, who is not involved in data collection or analysis, will be responsible for distributing the mouthguards to participants, ensuring that neither the principal investigator nor the participants know which type of mouthguard is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed custom-made mouth guards (Experimental): This arm will include participants receiving 3D printed custom mouth guards
  Interventions: Device: 3D printed custom-made mouth guards
- Traditional custom-made mouthguards (Active Comparator): Participants in the second group will receive traditional custom-made mouth guards
  Interventions: Device: Traditional custom-made mouth guards

INTERVENTIONS:
Device: 3D printed custom-made mouth guards — Participants in the first group will receive 3D printed custom-made mouth guards
  Arms: 3D printed custom-made mouth guards
Device: Traditional custom-made mouth guards — Participants in the active comparator arm will receive traditional custom-made mouth guards as an intervention
  Arms: Traditional custom-made mouthguards

SUMMARY:
This study aims to compare changes in the thickness of traditional and 3D-printed custom mouth guards in pediatric athletes who participate in contact sports. Specifically, it will assess the occlusal thickness changes between both types of mouth guards. The research will involve 56 children engaged in contact sports, and the evaluation will cover occlusal thickness, speech, oral functions, and cost-effectiveness over the course of one yea

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Cairo International Stadium, involving healthy children aged 8 to 14 who actively participate in contact sports and require mouthguards for safety. Participants must be physically fit and cooperative. With parental consent, they will be randomly assigned in a 1:1 ratio to one of two groups:

Group 1: Receives traditional custom-made mouthguards made from alginate impressions.

Group 2: Receives 3D-printed custom-made mouthguards created using digital intraoral scans and CAD/CAM 3D printing technology.

Primary Outcome: Changes in occlusal thickness will be measured at specific reference points on the occlusal surface using an Iwanson caliper. Measurements will be taken at baseline and again after 3 months.(7. Rossi, G. D., Lisman, P., & Leyte-Vidal, M. A. (2007))

Secondary Outcomes:

Knowledge, attitudes, and practices (KAP) related to mouthguard use, assessed via a structured questionnaire (Vignesh et al., 2023).

Cost-efficiency, evaluated using the incremental cost-effectiveness ratio (ICER).

after one year. Changes in oral functions and speech, measured with a validated Likert-scale questionnaire (Mat Zainal et al., 2024), administered at baseline, 3 months, and 6 months.

The trial aims to assess whether 3D-printed mouthguards offer equal or better protection against orofacial injuries compared to traditional mouthguards

ELIGIBILITY:
Inclusion Criteria:

Athletic children who play contact sports Age ranges between 8-14 years. Compliance: participants must agree to use mouth guard consistently Parental consent Physically fit

Exclusion Criteria:

Athletic children who play contact sports Age ranges between 8-14 years. Compliance: participants must agree to use mouth guard consistently Parental consent Physically fit

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Occlusal thickness changes | Three months
  This study will assess the wear patterns of both types of mouth guards in children participating in contact sports. The wear patterns will be measured by evaluating the thickness changes of the mouth guards over time using an Iwanson caliper (measured in millimeters, mm). This method will provide quantitative data on the durability and wear resistance of each type of mouth guard, helping to determine which type maintains its protective properties longer under the stress of regular use. The mouth guard thickness will be measured at two distinct time points (baseline and three months)

SECONDARY OUTCOMES:
Cost Efficiency of both mouth guards | One year
  This study will also assess the cost efficiency of both types of custom-made mouth guards by calculating the cost per unit, using the U.S Dollar (USD) as the unit of measurement. The incremental cost effectiveness ratio will be calculated after one year. The following equation will be used to measure the incremental cost-effectiveness ratio (Sadatsafavi et al., 2009): ICER=(Mouth guard A cost- Mouth guard B cost)/(outcome of mouth guard A-Outcome of mouth guard B)
Changes Speech and in Oral Functions | Six months
  Oral functions, such as speaking difficulty, lisping, nausea, bulkiness, and mouth dryness, will be evaluated using a validated questionnaire adapted from the study by Mat Zainal et al. (2024). This questionnaire will be administered at three separate time points: baseline, 3 months, and 6 months.
Knowledge, attitude, and practice (KAP) of children toward mouthguards | Initial visit
  The study will assess the knowledge, attitudes, and practices (KAP) of children regarding mouth guard use for preventing orofacial injuries during contact sports. It will focus on their awareness of the risks associated with orofacial injuries, their understanding of mouth guards as a protective tool, and their current usage habits. A structured questionnaire, adapted from Vignesh et al. (2023), will be administered to all participants in both groups during the initial visit.

CONTACTS AND LOCATIONS:
Overall Officials: Gihan Mohamed Abuelniel, Doctoral Degree (Professor), Study Director — Cairo University; Passant Nagi, Master's Degree, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be shared with qualified researchers upon request, following ethical guidelines and approval from the relevant ethics committee. The data will be anonymized to ensure participant confidentiality and will be made available through a secure data repository.

REFERENCES:
- [Background] Abbott PV, Tewari N, O'Connell AC, Mills SC, Stasiuk H, Roettger M, Levin L. The International Association of Dental Traumatology (IADT) and the Academy for Sports Dentistry (ASD) guidelines for prevention of traumatic dental injuries: Part 3: Mouthguards for the prevention of dental and oral trauma. Dent Traumatol. 2024 Feb;40 Suppl 1:7-9. doi: 10.1111/edt.12925. PMID 38363704
- [Background] Mat Zainal MK, Liew AKC, Abdullah D, Soo E, Abdul Hamid B, Ramlee RAM. Changes in oral functions and speech when using custom-fitted mouthguards: An uncontrolled before-and-after study. Dent Traumatol. 2024 Aug;40(4):460-469. doi: 10.1111/edt.12939. Epub 2024 Mar 8. PMID 38459669
- [Background] Singh G, Garg S, Damle SG, Dhindsa A, Kaur A, Singla S. A study of sports related occurrence of traumatic orodental injuries and associated risk factors in high school students in north India. Asian J Sports Med. 2014 Sep;5(3):e22766. doi: 10.5812/asjsm.22766. Epub 2014 Aug 28. PMID 25520762
- [Background] Tanaka Y, Maeda Y, Yang TC, Ando T, Tauchi Y, Miyanaga H. Prevention of orofacial injury via the use of mouthguards among young male rugby players. Int J Sports Med. 2015 Mar;36(3):254-61. doi: 10.1055/s-0034-1390498. Epub 2014 Oct 20. PMID 25329428
- [Background] Avgerinos S, Stamos A, Nanussi A, Engels-Deutsch M, Cantamessa S, Dartevelle JL, Unamuno E, Del Grosso F, Fritsch T, Crouzette T, Striegel M, Sanchez CC, Okshah A, Tzimpoulas N, Naka O, Kouveliotis G, Tzoutzas I, Zoidis P, Synodinos F, Loizos E, Tasopoulos T, Haughey J, Rahiotis C. Position Statement and Recommendations for Custom-Made Sport Mouthguards. Dent Traumatol. 2025 Jun;41(3):246-251. doi: 10.1111/edt.13019. Epub 2024 Nov 22. PMID 39578680
- [Background] Sadatsafavi M, Marra CA, Ayas NT, Stradling J, Fleetham J. Cost-effectiveness of oral appliances in the treatment of obstructive sleep apnoea-hypopnoea. Sleep Breath. 2009 Aug;13(3):241-52. doi: 10.1007/s11325-009-0248-4. Epub 2009 Feb 20. PMID 19229577